CLINICAL TRIAL: NCT04741594
Title: Alveolar Ridge Expansion by Osseodensification and Its Impact on Implant Survival and Success: A Case Series
Brief Title: Osseodensification and Implant Survival and Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12966
Record Dates: First submitted 2021-01-15; First posted 2021-02-05 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Missing Teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Versah group (Experimental)
  Interventions: Device: Densah

INTERVENTIONS:
Device: Densah — Alveolar bone remodeling after tooth extraction may result in significant ridge resorption and inadequate bone volume for implant placement. Several methods have been designed for ridge augmentation, among which is the new technique of osseodensification, using the Densah® burs by Versah® (Versah®, LLC, Jackson, MI, USA). This method compresses the trabecular bone to periphery of the osteotomy site and has shown up to 80% ridge expansion in animal histological studies , , , , , . Apart from being an animal model with a short follow-up, another limitation of these studies is the lack of three-dimensional evaluation of the change in morphology of the ridge. Human clinical studies , , , , have reported similar results, but they do not evaluate if this bone volume is retained during osseointegration and loading periods. No standardization method or long-term evaluation of peri-implant health was reported.

SUMMARY:
Approximately 40 implants from patients seeking treatment at the University of Oklahoma, College of Dentistry will be recruited for this study. Osteotomies will be prepared using the osseodensification technique and implants will be placed immediately after. The implants will be from a single manufacturer (Roxolid® SLA® Bone Level Tapered; Straumann®, Institut Straumann AG, Basel, Switzerland). Volumetric analysis of alveolar ridge will be studied using intra-surgical direct measurements and CBCT imaging. A custom stent will be fabricated to standardize the clinical and radiographic measurements at 2mm, 3mm, and 4mm apical to the alveolar crest. Changes in peri-implant bone density will be analyzed on standardized periapical and bitewing radiographs, using the ImageJ software (National Institute of Health, Bethesda, Maryland, USA). Implant stability quotient (ISQ) values will be recorded with a resonance frequency analysis system (Osstell®, Gothenburg, Sweden). Calibrated examiners will assess implant survival and biological or restorative complications and failures. Sites will be evaluated throughout osseointegration and one year after final restoration is delivered.

ELIGIBILITY:
4. Inclusion / Exclusion Criteria

The inclusion criteria include:

1. Adult patients ≥18 years old
2. Able to understand and sign a written informed consent form and willing to fulfil all study requirements
3. Healed edentulous ridge that is planned for an implant restoration.
4. Experimental site has not been previously augmented with xenograft
5. Experimental site has at least 2 mm of cancellous bone

The exclusion criteria include:

1. Uncontrolled systemic disease
2. Currently smoking >10 cigarettes/day
3. History of head/neck radiotherapy within the past five years
4. Current use of oral bisphosphonates or history of IV bisphosphonate use
5. Pregnant, expecting to become pregnant, or lactating women
6. Presence of active periodontal disease
7. Poor oral hygiene
8. Previous history of implant failure at the site

The early termination criteria include:

1. The researcher believes that it is not in the patient's best interest to stay in the study
2. Based on the exclusion criteria, the patient becomes ineligible to participate
3. Patient's medical condition requires interventions which preclude involvement in the study (radiation therapy, chemotherapy, etc)
4. Patient does not follow study related instructions
5. The study is suspended or canceled

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Bone width (mm) | 2 years
  Bone width at 2, 3, 4 mm apical to edentulous alveolar ridge.

SECONDARY OUTCOMES:
implant stability | 2 years
  Implant stability quotient (ISQ) values
Survival and failure rate | 2 years
  Rates of survival and failure rate

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, OUHSC, Oklahoma City, Oklahoma, United States